CLINICAL TRIAL: NCT07385742
Title: A Comparative Study Between Botulinum Toxin Versus Platelet Rich Fibrin Injection for Treatment of Temporomandibular Joint Internal Derangement
Brief Title: Botulinum Toxin Versus Platelet Rich Fibrin for TMJ Internal Derangement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 715/2023
Record Dates: First submitted 2026-01-25; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Temporomandibular Joint Internal Derangement; Temporomandibular Joint Disorders; Temporomandibular Disorders (TMD); TMJ Pain
Keywords: Temporomandibular Joint; TMJ Internal Derangement; Botulinum Toxin Type A; BOTOX Injection; Platelet Rich Fibrin; Injectable PRF; Lateral Pterygoid Muscle
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — proliferation regulatory factors, human urine; Injections; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: This study used a parallel assignment design in which 20 patients with temporomandibular joint internal derangement were randomly assigned into two equal groups. Group I received intracapsular injectable platelet-rich fibrin (I-PRF) into the superior joint space of the temporomandibular joint, while group II received botulinum toxin type A injections into the lateral pterygoid muscle. Each participant received only one of the two interventions and was followed for clinical and radiographic outcomes at one, three, and six months. The interventions were administered concurrently across groups, and the effects of each treatment were compared between the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-PRF Injection Group (Group I) (Experimental): This arm included 10 patients who underwent arthrocentesis of the temporomandibular joint, followed by 1 mL of intra-articular injectable platelet-rich fibrin (I-PRF).
  Interventions: Procedure: Injectable Platelet-Rich Fibrin (I-PRF) Injection
- Botulinum Toxin Injection Group (Group II) (Experimental): This arm included 10 patients who received an ultrasound-guided injection of 7 mL containing 35 units of botulinum toxin type A (BOTOX) into the lateral pterygoid muscle.
  Interventions: Drug: Botulinum Toxin Type A (BOTOX) Injection

INTERVENTIONS:
Procedure: Injectable Platelet-Rich Fibrin (I-PRF) Injection — Participants in this arm underwent arthrocentesis of the temporomandibular joint, followed by injection of 1 mL of intra-articular injectable platelet-rich fibrin (I-PRF) into the superior joint space.
  Other Names: I-PRF; Autologous Platelet-Rich Fibrin
  Arms: I-PRF Injection Group (Group I)
Drug: Botulinum Toxin Type A (BOTOX) Injection — Participants in this arm received an ultrasound-guided injection of 7 mL containing 35 units of botulinum toxin type A (BOTOX) into the lateral pterygoid muscle.
  Other Names: BTX-A; Botulinum Neurotoxin Type A
  Arms: Botulinum Toxin Injection Group (Group II)

SUMMARY:
Temporomandibular joint (TMJ) internal derangement is a common cause of temporomandibular disorders and is often associated with pain, restricted mandibular movement, joint sounds, and functional limitations during mastication and mouth opening. Various treatment modalities have been proposed to manage these symptoms, aiming to reduce pain and improve joint function.

This randomized clinical study was conducted to compare the effectiveness of botulinum toxin type A (BOTOX) injection into the lateral pterygoid muscle versus intracapsular injection of injectable platelet-rich fibrin (I-PRF) in the management of TMJ internal derangement. A total of 20 patients diagnosed with TMJ internal derangement were randomly allocated into two equal groups. Group I received intracapsular I-PRF injections into the superior joint space of the temporomandibular joint, while group II received botulinum toxin injections into the lateral pterygoid muscle.

Clinical evaluation was performed using subjective and objective parameters at one, three, and six months following treatment. Outcomes included assessment of pain, maximum mouth opening, mandibular movements, joint tenderness, and muscle tenderness upon palpation. Radiographic evaluation was conducted using magnetic resonance imaging (MRI) to assess intra-articular changes of the temporomandibular joint following the interventions.

The study aimed to determine which treatment modality provided superior clinical and radiographic outcomes for the management of TMJ internal derangement.

DETAILED DESCRIPTION:
Temporomandibular joint (TMJ) internal derangement represents a common cause of temporomandibular disorders (TMDs) and is frequently associated with pain and functional limitations. Patients affected by TMJ internal derangement commonly present with pain during mastication, difficulty or pain during mouth opening, joint sounds such as clicking or crepitation, and preauricular pain. Due to the multifactorial nature of this condition, numerous treatment modalities have been investigated to achieve effective symptom relief and functional improvement.

The aim of this clinical study was to evaluate and compare the effectiveness of botulinum toxin type A (BOTOX) injection into the lateral pterygoid muscle versus intracapsular injection of injectable platelet-rich fibrin (I-PRF) for the management of TMJ internal derangement.

This randomized clinical study was conducted on a total of 20 patients diagnosed with TMJ internal derangement. The participants were randomly and equally allocated into two groups using an online randomization tool (www.randomizer.org). Group I consisted of 10 patients who received intracapsular injections of injectable platelet-rich fibrin (I-PRF) into the superior joint space of the temporomandibular joint. Group II consisted of 10 patients who received botulinum toxin type A injections into the lateral pterygoid muscle.

Patients in both groups were evaluated using both subjective and objective parameters at baseline and during follow-up periods at one month, three months, and six months following injection. Clinical evaluation included assessment of pain, maximum mouth opening, and mandibular movements in all directions to determine improvement in mouth mobility. Tenderness was assessed by palpation of the masticatory muscles, including the temporalis, masseter, and lateral pterygoid muscles, as well as palpation of the temporomandibular joint through the external auditory canal.

Radiographic evaluation was performed using magnetic resonance imaging (MRI) to assess intra-articular changes of the temporomandibular joint following treatment. MRI findings were used to evaluate joint structure, disc position, and overall intra-articular condition after the intervention.

The outcomes of this study were analyzed to determine which treatment modality provided superior clinical and radiographic improvement in patients with TMJ internal derangement.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15 to 50 years.
* Adults of both genders.
* Patients free from systemic disease (ASA I).
* Patients presenting with persistent symptoms and signs of temporomandibular disorders, specifically anterior disc displacement with reduction (ADDwR).
* Patients willing to comply with the follow-up schedule and treatment protocol.

Exclusion Criteria:

* Pregnant or lactating women, or women with osteoporosis.
* Patients who have had previous TMJ surgery.
* Patients who have undergone previous arthrocentesis.
* Any other temporomandibular joint disease that may confound diagnosis (e.g., myofascial pain-dysfunction syndrome, MPDS).
* Patients allergic to components of the injection solutions.
* Patients with previous trauma to the TMJ.
* Patients with metal bullets in the body, metallic foreign body in the eye, or intracranial aneurysm clips (unless made of titanium).
* Patients using anticoagulant or immunosuppressive medications.

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-04-19 (Actual)

PRIMARY OUTCOMES:
Pain Score (Visual Analogue Scale, VAS) | 1 month, 3 months, and 6 months post-injection
  Pain associated with temporomandibular joint internal derangement was assessed using a 10-point visual analogue scale (VAS), where 0 indicates no pain and 10 indicates the worst pain. Pain was measured at baseline (pre-injection) and at follow-up visits. Comparisons were made within each group over time and between the I-PRF and BOTOX groups to determine the relative effectiveness of each treatment in reducing TMJ pain.
Joint Sounds (Clicking) Assessment | 1 month, 3 months, and 6 months post-injection
  The presence or absence of TMJ clicking was assessed by bimanual palpation during mouth opening and closing. Changes over time were recorded within groups and between the I-PRF and BOTOX groups.
MRI Assessment of Disc Position | Baseline, 1 month, 3 months, and 6 months post-injection
  MRI was performed to evaluate the position and structure of the TMJ articular disc. Disc positions were categorized as Superior (Normal), Reducing Disc Displacement (RDD), or Non-Reducing Disc Displacement (NRDD). Changes were compared within each group over time and between groups.

SECONDARY OUTCOMES:
Maximal Mouth Opening (MMO) | 1 month, 3 months, and 6 months post-injection
  MMO was measured from the incisal edge of the upper central incisors to the incisal edge of the lower central incisors using a digital caliper. Measurements were taken at baseline and follow-up visits. Changes were compared within and between the I-PRF and BOTOX groups to evaluate improvement in mouth opening.
Lateral Mandibular Movements (Right and Left) | 1 month, 3 months, and 6 months post-injection
  Right and left lateral mandibular movements were measured from the maxillary midline using a millimeter ruler or caliper. Changes in lateral movement were evaluated within each group over time and between groups.
Protrusive Mandibular Movement (PM) | 1 month, 3 months, and 6 months post-injection
  Protrusive mandibular movement was measured from the midpoint of the maxillary central incisors to the midpoint of the mandibular central incisors using a millimeter ruler or caliper. Progression was assessed within each group and between the I-PRF and BOTOX groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Said Hamed, Professor, Study Chair — Professor of Oral and Maxillofacial Surgery, Faculty of Dentistry - Suez Canal University; Ahmed Abd elmohsen Younis, Assistant. Professor, Study Director — Assistant. Professor of Oral and Maxillofacial Surgery, Faculty of Dentistry - Suez Canal University
Locations (1):
- Suez Canal University, Faculty of Dentistry, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoshida K. Botulinum Neurotoxin Injection for the Treatment of Recurrent Temporomandibular Joint Dislocation with and without Neurogenic Muscular Hyperactivity. Toxins (Basel). 2018 Apr 25;10(5):174. doi: 10.3390/toxins10050174. PMID 29693593
- [Background] George SJ, Boscoe MJ. Inhaled nitric oxide for right ventricular dysfunction following cardiac transplantation. Br J Clin Pract. 1997 Jan-Feb;51(1):53-5. PMID 9158275
- [Background] Manafikhi M, Ataya J, Heshmeh O. Evaluation of the efficacy of platelet rich fibrin (I-PRF) intra-articular injections in the management of internal derangements of temporomandibular joints - a controlled preliminary prospective clinical study. BMC Musculoskelet Disord. 2022 May 14;23(1):454. doi: 10.1186/s12891-022-05421-7. PMID 35568935
- [Background] Chung PY, Lin MT, Chang HP. Effectiveness of platelet-rich plasma injection in patients with temporomandibular joint osteoarthritis: a systematic review and meta-analysis of randomized controlled trials. Oral Surg Oral Med Oral Pathol Oral Radiol. 2019 Feb;127(2):106-116. doi: 10.1016/j.oooo.2018.09.003. Epub 2018 Sep 26. PMID 30449691
- [Background] Bousnaki M, Bakopoulou A, Koidis P. Platelet-rich plasma for the therapeutic management of temporomandibular joint disorders: a systematic review. Int J Oral Maxillofac Surg. 2018 Feb;47(2):188-198. doi: 10.1016/j.ijom.2017.09.014. Epub 2017 Oct 20. PMID 29066000
- [Background] Bakke M, Moller E, Werdelin LM, Dalager T, Kitai N, Kreiborg S. Treatment of severe temporomandibular joint clicking with botulinum toxin in the lateral pterygoid muscle in two cases of anterior disc displacement. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Dec;100(6):693-700. doi: 10.1016/j.tripleo.2004.11.019. PMID 16301150
- [Background] Albilia J DMD, MSc, Herrera-Vizcaino C DDS, Weisleder H BSc, Choukroun J MD, Ghanaati S MD, DMD, PhD. Liquid platelet-rich fibrin injections as a treatment adjunct for painful temporomandibular joints: preliminary results. Cranio. 2020 Sep;38(5):292-304. doi: 10.1080/08869634.2018.1516183. Epub 2018 Sep 20. PMID 30231809